CLINICAL TRIAL: NCT02812108
Title: Investigation of Clinical and Hemodynamic Factors Affecting the Outcome of Intracranial Aneurysm Embolization
Brief Title: Hemodynamic Analysis for Intracranial Aneurysms Recanalization After Endovascular Treatment
Acronym: HARET
Status: Completed | Type: Observational
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Principal Investigator, Xinjian Yang, MD, Vice Chair of Department of Interventional Neuroradiology, Beijing Neurosurgical Institute
Other Study IDs: NSFC-81220108007
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Intracranial Aneurysm
Keywords: intracranial aneurysm; endovascular treatment; recanalization; outcome; hemodynamics; computational fluid dynamic; stent; flow diversion
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood

GROUPS / COHORTS (1):
- HARET: All patients with intracranial aneurysms, ruptured or unruptured, treated by endovascular treatment
  Interventions: Device: intracranial stent, flow diverter and coils

INTERVENTIONS:
Device: intracranial stent, flow diverter and coils
  Other Names: Low profile Visualized Intraluminal Device (LVIS);; Pipeline™(or Flex) Embolization Device;

SUMMARY:
This study was designed to collect a large series of patients with aneurysms treated endovascularly to analyze hemodynamic factors that affect aneurysm recanalization.

DETAILED DESCRIPTION:
With the rapid development of endovascular technique, endovascular treatment has become the first line treatment for intracranial aneurysms (IAs). Compared to microsurgical clipping, less invasive and lower morbidity have been shown after endovascular treatment. However, the aneurysms recanalization is the drawback of such modality. It has been reported that many factors, including complete initial embolization, stent assisted coiling, dense packing and flow diverter, could reduce recanalization rate. Larger size, wide neck, rupture status and intraluminal thrombosis are reported as risk factors of aneurysm recanalization. However, no analysis of hemodynamic risk factors affecting the aneurysm recanalization has been conducted in a large prospective series of patients.

Hemodynamics is reported to play an important role in aneurysm initiation, growth and rupture. Previous studies have showed that the hemodynamics is associated with outcomes of aneurysms after endovascular treatment. High wall shear stress and flow velocity are risk factors of aneurysm recanalization. However, the relationship between hemodynamics and aneurysm outcomes is still unclear. To explore the hemodynamic predictors of aneurysm recanalization is of great value for clinical practice.

Hemodynamic analysis for intracranial aneurysms recanalization after endovascular treatment (HARET) is a prospective trial designed to collect a large series of patients with aneurysms treated endovascularly to analyze hemodynamic factors that affect aneurysm recanalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by endovascular approach for intracranial aneurysm(s)
* Patients older than 18 years
* Patients accepting to participate to the study

Exclusion Criteria:

* Patients already treated by endovascular approach for an intracranial aneurysm
* Patients having a brain arteriovenous malformation
* Patients having a fusiform aneurysm
* Patients having a dissecting aneurysm
* Patients treated by parent vessel occlusion
* Patients treated by covered stent
* Patients lacking 3-dimensional aneurysm images or the images not satisfied the simulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with intracranial aneurysms, ruptured or unruptured, treated by endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
hemodynamic factors related to aneurysm recanalization as assessed by computational blood flow simulation | assessed at 6 months (plus or minus 3 months) after procedure
  Using computational fluid dynamic method, the parameters as wall shear stress (WSS), flow velocity, pressure could be calculated and analyzed. These will be studied as a composite indicator for recanalization assessment.

SECONDARY OUTCOMES:
clinical factors related to aneurysm recanalization as recorded from medical chart | assessed at 6 months (plus or minus 3 months) after procedure
  for clinical risk factors as aneurysm size, neck size, treatment method, device use, follow-up interval, smoke history, hypertension, et al, will be recorded and analyzed.These will be studied as a composite indicator for recanalization assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Neurosurgical Institute and Beijing Tiantan Hospital, Beijing, China

REFERENCES:
- [Derived] Liu J, Zhang Y, Wang A, Zhang Y, Li Y, Yang X. Haemodynamic analysis for recanalisation of intracranial aneurysms after endovascular treatment: an observational registry study in China. BMJ Open. 2017 May 12;7(5):e014261. doi: 10.1136/bmjopen-2016-014261. PMID 28501811